CLINICAL TRIAL: NCT02836925
Title: A Multicenter Study to Evaluate the Anti-viral Activity of an Interferon-free Treatment With Ledipasvir/Sofosbuvir (G1 and G4) and Sofosbuvir/Velpatasvir (G2 and G3) for Patients With Hepatitis C Virus-associated Indolent B-cell Lymphomas
Brief Title: Ledipasvir+Sofosbuvir and Sofosbuvir+Velpatasvir for Pts With Indolent Bcell Lymphoma Associated With HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_BArT
Record Dates: First submitted 2016-02-25; First posted 2016-07-19 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Indolent B-cell Lymphoma; Hepatitis C
Keywords: hepatitis C; NHL; Indolent B-cell lymphoma
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ledipasvir+Sofosbuvir,Sofosbuvir+Velpatasvir (Experimental): The study includes an antiviral treatment with interferon-free regimen followed by lymphoma restaging; following the end of antiviral treatment patients will be evaluated for sustained virological response and safety parameters every 3 months for 1 year and then every 6 months for 2 years. ORR and vital status will be also evaluated
  Interventions: Drug: Ledipasvir+Sofosbuvir; Drug: Sofosbuvir+Velpatasvir

INTERVENTIONS:
Drug: Ledipasvir+Sofosbuvir — Patients with genotype 1 or genotype 4 Ledipasvir 90 mg + Sofosbuvir 400 mg
  * 12 weeks in previously untreated infected patients
  * 24 weeks for previously treated patients with uncertain subsequent retreatment options
  Other Names: Harvoni
Drug: Sofosbuvir+Velpatasvir — Patients with genotype 2 or genotype 3 Sofosbuvir 400 mg + Velpatasvir 100 mg
  · 12 weeks of treatment
  Other Names: Epclusa

SUMMARY:
This is a non-randomized, a single arm, phase II multicentre study of sofosbuvir plus ledipasvir (genotype 1 and 4) or sofosbuvir plus velpatasvir (genotype 2 and 3) for patients with hepatitis C virus-associated indolent B-cell lymphomas (HCV-RNA positive).

DETAILED DESCRIPTION:
The study includes an antiviral treatment with interferon-free regimen followed by lymphoma restaging; following the end of antiviral treatment patients will be evaluated for sustained virological response and safety parameters every 3 months for 1 year and then every 6 months for 2 years. ORR and vital status will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Indolent B cell lymphoma including: marginal zone lymphoma (nodal, extranodal, splenic and disseminated), lymphoplasmacytic lymphoma, small lymphocytic lymphoma, follicular lymphoma grade 1 and 2, CD5-negative B-cell lymphoma NOS
3. HCV-RNA positivity
4. Assessable HCV genotype
5. No previous therapy for the lymphoma
6. Measurable disease after diagnostic biopsy (longest axis ≥1.5 cm for nodal and ≥1 cm for extranodal lesions) and/or evaluable disease (quantifiable BM infiltrate and ≥5 x 109/l clonal B-cell in peripheral blood in case of exclusive BM/leukemic disease in CD5-negative Bcell lymphoma NOS)
7. No need of immediate lymphoma treatment defined as absence of all the following criteria: systemic symptoms, bulky nodal or extranodal mass (>7 cm), symptomatic splenomegaly, progressive leukemic phase, serous effusions
8. Performance status <2 according to ECOG scale
9. Adequate hematological counts: ANC >1 x 109/L, hemoglobin >9 g/dl (transfusion independent), platelet count > 50 x 109/L (transfusion independent)
10. No central nervous system (CNS) disease (meningeal and/or brain involvement by lymphoma)
11. Adequate kidney function (creatinine clearance ≥ 45 ml/min)
12. Cardiac ejection fraction ≥45% (echocardiography or MUGA scan)
13. Normal lung function
14. Non peripheral neuropathy or active neurological non neoplastic disease of CNS
15. Non major surgical intervention prior 3 months to enrolment if not due to lymphoma and/or no other disease life-threatening that can compromise chemotherapy treatment
16. Disease free of prior malignancies other than lymphoma for >3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
17. Life expectancy > 6 months
18. No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
19. Written informed consent
20. Women must be:

    * postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
    * surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
    * completely abstinent (at the discretion of the investigator/per local regulations) (periodic abstinence from intercourse is not permitted) or
    * if sexually active, be practicing a highly effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (eg: condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, before entry, and must agree to continue to use the same method of contraception throughout the study. They must also be prepared to continue birth control measures for at least 6 months after terminating treatment.
21. Women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening
22. Men must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study. Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 1 month after receiving the last dose of study drug if not taking ribavirin of for 6 months after receiving the last dose of study drug if taking ribavirin.

Exclusion Criteria:

1. Diagnosis of lymphoblastic lymphoma, Burkitt lymphoma, diffuse large B-cell lymphoma, mantle cell lymphoma, follicular lymphoma grade 3, primary mediastinal B-cell lymphoma
2. Previous anti-HCV treatment with sustained virological response
3. Diagnosis of cirrhosis (histological or Stiffness >12 KpA)
4. CNS disease (meningeal and/or brain involvement by lymphoma)
5. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
6. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug)
7. Concomitant therapy with amiodarone
8. Uncontrolled or severe cardiovascular disease including myocardial infarction within six months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina,
9. Cardiac ejection fraction <45% (MUGA scan or echocardiography).
10. Creatinine clearance <45 ml/min
11. Presence of major neurological disorders
12. HIV positivity, HBV positivity (HbsAg+ or HBV-DNA+) with the exception of HBcAb+, HbsAg-, HBsAb+/- patients with HBV-DNA negativity
13. Ongoing systemic bacterial, fungal or viral infections at the time of initiation of study treatment (defined as requiring therapeutic dosing of an antimicrobial, antifungal or antiviral agent)
14. Major surgical intervention prior 3 months to enrollment if not due to lymphoma and/or other
15. Prior malignancies other than lymphoma in the last 3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
16. Life expectancy <6 months
17. Any other coexisting medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
18. If female, the patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2020-02 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
SVR12 | 12 weeks from the end of the treatment
  Sustained virologic response (SVR12) defined as undetectability of HCV-RNA 12 weeks after completion of antiviral therapy

SECONDARY OUTCOMES:
ORR | 12 weeks from the end of treatment
  Overall response rate (ORR) of lymphoma: CR is defined by the complete disappearance of all detectable sites and symptoms; PR is defined as a more than 50% reduction. Responses different from CR/PR are defined as stable disease (SD); progressive disease (PD) is considered an increase in size of more than 50% of previously documented disease or the appearance of new lesions. Lymphoma response will be assessed 12 weeks after the end of antiviral treatment
PFS | 36 months
  Progression-free survival (PFS) defined as the time between enrolment and progression or relapse or death from any cause.
EFS | 36 months
  Event-free survival (EFS) defined as time between enrolment and failure of treatment or death as a result of any cause
OS | 36 months
  Overall survival (OS) defined as the time between enrolment and death from any cause
ORR for lymphoma | 12 weeks from the end of treatment
  ORR for lymphoma according to Matutes criteria (Matutes et al, Leukemia 2008) only in patients with splenic-marginal zone lymphoma (SMZL)
Rapid virological response | 4 weeks
  rapid virologic response (RVR)
Extended rapid virological response | 4 weeks
  extended RVR (eRVR)
Early virological response | 4 weeks
  early virologic response (EVR)
Toxicity - Incidence of Adverse Events | 12 months
  toxicity will be classified according to definitions of Common Terminology Criteria for Adverse Event version 4.03 (CTCAE). It will be determined by the incidence of severe, life-threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Luca Arcaini, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (13):
- Italy (13):
  - A.O. Spedali Civili, Brescia, BS
  - Irccs Centro Di Riferimento Oncologico (Cro), Aviano, Pordenone
  - Ospedale San Bortolo, Vicenza, VI
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele Ematologia, Milan
  - U.O. Ematologia AO di Padova, Padua
  - A.O. Universitaria Di Parma, Parma
  - Ematologia Policlinico San Matteo, Pavia
  - Ospedale Civile Piacenza, Piacenza
  - Ematologia - Policlinico Umberto I Università Sapienza, Roma
  - Dipartimento di Oncologia Medica ed Ematologia, Istituto Humanitas, Rozzano
  - AOU Città della Salute e della Scienza di Torino, Torino
  - Ospedale di Circolo e Fondazione Macchi, Varese

REFERENCES:
- [Derived] Merli M, Rattotti S, Spina M, Re F, Motta M, Piazza F, Orsucci L, Ferreri AJM, Perbellini O, Dodero A, Vallisa D, Pulsoni A, Santoro A, Sacchi P, Zuccaro V, Chimienti E, Russo F, Visco C, Zignego AL, Marcheselli L, Passamonti F, Luminari S, Paulli M, Bruno R, Arcaini L; Fondazione Italiana Linfomi. Direct-Acting Antivirals as Primary Treatment for Hepatitis C Virus-Associated Indolent Non-Hodgkin Lymphomas: The BArT Study of the Fondazione Italiana Linfomi. J Clin Oncol. 2022 Dec 10;40(35):4060-4070. doi: 10.1200/JCO.22.00668. Epub 2022 Jun 17. PMID 35714311